CLINICAL TRIAL: NCT04519463
Title: The Effect of Local Anesthesia With Lidocaine During Insertion and Removal of Nasal Packing
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Muhamed Masalha (Other)
Responsible Party: Sponsor-Investigator, Muhamed Masalha, Dr, Muhamed Masalha; Principal Investigator; Senior Surgeon in the Endoscopic Sinus Surgery Unit, the Department of Otolaryngology-Head and neck surgery, HaEmek Medical Center, Israel
Organization: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0081-20-EMC
Record Dates: First submitted 2020-08-06; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Epistaxis; Analgesia
Keywords: Nasal Spray; Nasal Anesthesia; Epistaxis
MeSH Terms: conditions — Epistaxis; Agnosia

STUDY DESIGN:
Intervention Model Description: Double-Blind Randomized Controlled Trial
Who Masked: Participant, Investigator
Masking Description: Both Xylocaine spray and Placebo (saline) will be in similar containers with serial numbers, Both clinician and patient are blinded to the content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Xylocaine (Experimental): 30 patients who receive Xylocaine 10% nasal spray
  Interventions: Drug: Xylocaine Mucosal Product
- Saline (Placebo Comparator): 30 patients who receive saline nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xylocaine Mucosal Product — Xylocaine 10% Nasal Spray
  Arms: Xylocaine
Drug: Placebo — Sodium Chloride 0.9%
  Arms: Saline

SUMMARY:
This study aims to investigate the effect of local nasal anesthesia with lidocaine spray on the insertion of nasal tampons during active nasal bleeding.

DETAILED DESCRIPTION:
Nasal packing has many uses, such as prevention of postoperative bleeding following endoscopic sinus surgery, stabilization of the nasal septum, prevention of adhesions following septoplasty, and treatment of active epistaxis1,2.

The utilization of tampons for nasal packing during nasal and sinus surgeries is widely used and safe. Nasal tampons assist in creating a moist supportive environment for tissue healing without causing local irritation or foreign body reaction3. The removal is performed after 24-48 hours. On the other hand, there are some disadvantages to the uses of nasal tampons: trauma to the nasal mucosa, infection of the nose and sinuses, aspiration of part of the tampon, and even toxic shock syndrome3. One of the most troublesome aspects to the patient and the clinician is the pain and discomfort during insertion and removal of the tampons3,4. In our experience, these symptoms are of considerable significance to the patient experience and satisfaction.

There is a wide range of commercially available nasal packings such as Merocel and Nasopore.

In our practice, Merocel nasal tampons are used, which contain polyvinyl acetate. This type of material expands upon contact with fluids, and it is not soluble. This product is used at the end of endoscopic nasal surgeries and in the treatment of active epistaxis, not amenable to local pressure and without a recognizable source of bleeding. In case of unstoppable bleeding despite the use of nasal tampons, a nasal balloon is inflated in the nasal cavity. Its insertion and inflation are associated with patient pain and discomfort.

Lidocaine is a drug commonly used for local anesthesia. It is used for local nasal anesthesia by a variety of commercially available sprays, atomizers, nebulizers, gels, and ointments. Lidocaine causes local anesthesia by affecting sodium channels, causing decreased initiation and conduction of neural impulses. In turn, fewer afferent impulses reach the central nervous system6. In healthy individuals, side effects are negligible, but it could influence patients with cardiac infarction. The main side effects of lidocaine are neurological, which could be of significance in the case of inflamed or damaged tissue because of rapid absorption. The use of Lidocaine spray (Xylocaine 10%) is commonly available worldwide and is routinely used in our institution before fiberoptic laryngoscopy.

Previous publications have mentioned the positive effect of local anesthesia during the removal of nasal tampons5,7. In a recent meta-analysis, local anesthetics were associated with less pain during the removal of nasal tampons and shortened time of the procedure. Yet, the authors recognized the need for additional randomized controlled trials7. There are no previous publications on the effect of local anesthetics on the insertions of nasal tampons during active nasal bleeding. In the experience of the senior author, for many years, the application of lidocaine spray 10% before the insertions of nasal tampons for epistaxis was associated with a significant reduction of pain and discomfort.

This study aims to investigate the effect of local nasal anesthesia with lidocaine spray on the insertion of nasal tampons during active nasal bleeding. Secondary objectives include the impact on nasal tampons removal after the cessation of nasal bleeding and after endoscopic sinus surgery.

Research hypothesis: local anesthesia with lidocaine before the insertion of nasal tampons or inflatable balloon reduces patients' pain, discomfort, and stress during insertion for the treatment of active nasal bleeding, and during removal of nasal tampons either postoperatively or after cessation of epistaxis.

The study population involves 30 patients with spontaneous epistaxis and another 30 patients who went tampon removal postoperatively in our institution. Recruitment includes patients who came to the emergency department with active epistaxis and still had active bleeding after the application of local pressure without an identified source of bleeding, requiring treatment with tampons or an inflatable balloon. The second group included patients who require postoperative removal of nasal tampons.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Both sexes
* No known allergy for local anesthetics agents
* Patients with active nasal bleeding requiring the insertion of a tampon or an inflatable balloon, or patients requiring tampon removal postoperatively.

Exclusion Criteria:

* Age under 18 years.
* Known allergy to local anesthetics
* Lack of willingness to participate in a clinical trial
* Patient unable to give informed consent from any reason
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Immediately after the procedure
  Visual Analogue Scale (VAS) ranging from 0- no pain at all to 10 - unbearable pain.

SECONDARY OUTCOMES:
Patient Questionnaires | Immediately after the procedure
  Patient symptoms: nausea, vomiting, allergic reaction, localized pain, numbness in the pharynx, bitter taste, dysphagia. For any side effect, the duration until the symptoms had passed. Scale of symptoms severity ranging from 0- no symptoms at all to 10 - worst symptoms severity.

CONTACTS AND LOCATIONS:
Overall Officials: Muhamed Masalha, MD, Principal Investigator — Emek Medical Center, Afula, Israel.
Locations (1):
- Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watson MG, Campbell JB, Shenoi PM. Nasal surgery: does the type of nasal pack influence the results? Rhinology. 1989 Jun;27(2):105-11. PMID 2781213
- [Background] Weber R, Keerl R, Hochapfel F, Draf W, Toffel PH. Packing in endonasal surgery. Am J Otolaryngol. 2001 Sep-Oct;22(5):306-20. doi: 10.1053/ajot.2001.26499. PMID 11562881
- [Background] Haytoglu S, Kuran G, Muluk NB, Arikan OK. Different anesthetic agents-soaked sinus packings on pain management after functional endoscopic sinus surgery: which is the most effective? Eur Arch Otorhinolaryngol. 2016 Jul;273(7):1769-77. doi: 10.1007/s00405-015-3807-2. Epub 2015 Oct 28. PMID 26511988
- [Background] Karaaslan K, Yilmaz F, Gulcu N, Yigit B, Kocoglu H. The effect of prilocaine and prilocaine plus meperidine infiltration on the pain during nasal packing removal. Rhinology. 2007 Dec;45(4):321-4. PMID 18085028
- [Background] Tsai SC, Lai MT, Kao YL, Wu CC. Effect of infiltrating nasal packing with local anesthetics in postoperative pain and anxiety following sinonasal surgeries: a systemic review and meta-analysis. Braz J Otorhinolaryngol. 2020 May-Jun;86(3):376-382. doi: 10.1016/j.bjorl.2019.12.011. Epub 2020 Feb 12. PMID 32127341
- See also: Lidocaine Drug Information — https://www.hamichlol.org.il/%D7%9C%D7%99%D7%93%D7%95%D7%A7%D7%90%D7%99%D7%9F